CLINICAL TRIAL: NCT07052370
Title: TCRαβ-depleted Progenitor Cell Graft With Early Memory T-cell DLI, Plus Selected Use of Blinatumomab, in naïve T-cell Depleted Haploidentical Donor Hematopoietic Cell Transplantation for Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAP3HCT; NCI-2025-04293 (Other: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Hematologic Malignancy
Keywords: Hematopoietic Cell Transplant
MeSH Terms: conditions — Hematologic Neoplasms | interventions — thymoglobulin; Cyclophosphamide; fludarabine; Thiotepa; Melphalan; Mesna; Filgrastim; blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- HAP3HCT Treatment (Experimental): Prior to the infusion of donor cells, a preparative regimen consisting of antibodies and chemotherapy will be given. The preparative regimen includes the following total dosages: ATG 5mg/kg (over days -12 to -10); Cyclophosphamide 60 mg/kg (day -9); Fludarabine 150 mg/m2 (over days -8 to -4); Thiotepa 10 mg/kg (divided in two doses on day -3); Melphalan 70 mg/m2 (over days -2 to -1). Following this regimen the TCRαβ-depleted haploidentical donor product will be given on day 0 (subsequent infusion given on day +1 if needed to achieve goal CD34+ cell dose. Approximately 2 weeks later the memory cell donor lymphocyte infusion (DLI) will be given at a dose previously determined to be safe and effective.
  Blinatumomab will be empirically added for patients with CD19+ malignancy and given at least four weeks after the memory cell DLI.
  Interventions: Drug: Thymoglobulin; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Thiotepa; Drug: Melphalan; Drug: Mesna; Drug: Filgrastim; Drug: Blinatumomab; Device: CliniMACS

INTERVENTIONS:
Drug: Thymoglobulin — IV
Drug: Cyclophosphamide — IV
Drug: Fludarabine — IV
Drug: Thiotepa — IV
Drug: Melphalan — IV
Drug: Mesna — IV
Drug: Filgrastim — IV
Drug: Blinatumomab — IV
Device: CliniMACS — The mechanism of action of the CliniMACS Cell Selection System is based on magnetic-activated cell sorting (MACS). The CliniMACS device is a powerful tool for the isolation of many cell types from heterogeneous cell mixtures, (e.g. apheresis products). These can then be separated in a magnetic field using an immunomagnetic label specific for the cell type of interest.

SUMMARY:
This is a phase I, prospective clinical trial studying the safety and feasibility of providing early memory T-cell DLI.

The primary objective is:

- To assess the safety and feasibility of early CD45RA-depleted DLI administration.

The secondary objectives are

* To assess the safety and feasibility of the addition of blinatumomab in the early post-transplant period in patients with CD19+ malignancy.
* To measure and describe the pharmacokinetics of rabbit ATG in HCT recipients on this study.

DETAILED DESCRIPTION:
The purpose of the study is to learn more about the effects (good and bad) of transplanting progenitor (blood making) cells and donor lymphocytes (white blood cells) donated by a partially matched family member that have been modified in a laboratory, to children and young adults with a high risk cancer that is in remission but is at high risk of relapse. This study builds upon what we have learned from recently completed studies and will be testing the safety and effects of the chemotherapy and the combination of two different types of blood cell infusions on the transplant recipient's disease and overall survival.

In this study, participants with high-risk hematologic malignancies who lack an available suitable human leukocyte antigen (HLA) matched related/sibling donor (MSD) or matched unrelated donor (MUD), will undergo allogeneic hematopoietic cell transplantation (HCT) consisting of a TCRαβ-depleted haploidentical donor product with additional memory cell donor lymphocyte infusion (DLI) given in the early postHCT time period.

Prior to the infusion of donor cells, a preparative regimen consisting of antibodies and chemotherapy will be given. The preparative regimen includes the following total dosages: ATG 5mg/kg (over days -12 to -10); Cyclophosphamide 60 mg/kg (day -9); Fludarabine 150 mg/m2 (over days -8 to -4); Thiotepa 10 mg/kg (divided in two doses on day -3); Melphalan 70 mg/m2 (over days -2 to -1). Following this regimen the TCRαβ-depleted haploidentical donor product will be given on day 0 (subsequent infusion given on day +1 if needed to achieve goal CD34+ cell dose. Approximately 2 weeks later the memory cell donor lymphocyte infusion (DLI) will be given at a dose previously determined to be safe and effective.

Blinatumomab will be empirically added for patients with CD19+ malignancy and given at least four weeks after the memory cell DLI.

ELIGIBILITY:
Inclusion Criteria:

Recipient:

* Age less than or equal to 21 years
* High risk hematologic malignancy whereas allogeneic transplantation is the current standard of care. This includes (but is not limited to):

  * High risk ALL in CR1 or CR2,
  * any ALL in CR3 or subsequent;
  * AML in high risk CR1 (AML diagnosis includes myeloid sarcoma),
  * any AML in CR2 or subsequent,
  * any therapy related AML;
  * MDS (primary or secondary),
  * NK cell, biphenotypic, or undifferentiated leukemia/lymphoma in CR1 or subsequent;
  * CML in accelerated phase, or in chronic phase with persistent molecular positivity or intolerance to tyrosine kinase inhibitor, or a history of blast crisis.
* If prior CNS leukemia, it must be treated and in CNS CR
* Left ventricular ejection fraction > 40%, or shortening fraction ≥ 25%
* Creatinine clearance (CrCl) or glomerular filtration rate (GFR) ≥ 50 ml/min/1.73m2
* Forced vital capacity (FVC) ≥ 50% of predicted value; or pulse oximetry ≥ 92% on room air if patient is unable to perform pulmonary function testing
* Karnofsky or Lansky (age dependent) performance score ≥ 50 (See APPENDIX A)
* Bilirubin ≤ 3 times the upper limit of normal for age
* Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) ≤ 5 times the upper limit of normal for age

Donor:

* At least single haplotype matched (≥ 4 of 8) family member
* At least 18 years of age
* HIV negative
* Regarding donation eligibility, is identified as either:

  * Completed the process of donor eligibility determination as outlined in 21 CFR 1271 and agency guidance; OR
  * Does not meet 21 CFR 1271 eligibility requirements, but has a declaration of urgent medical need completed by the principal investigator or physician sub-investigator per 21 CFR 1271

Exclusion Criteria:

Recipient:

* Has a suitable HLA-identical sibling or suitable 12/12 (HLA-A, B, C, DRB1, DQB1, and DPB1) HLA-matched unrelated donor available in an appropriate time frame.
* Any other active malignancy other than the one for which this HCT is indicated
* Received a prior allogeneic HCT at any time
* Received an autologous HCT within the previous 6 months
* Pregnant, if female is of childbearing potential, negative test must be confirmed by serum or urine pregnancy test within 14 days prior to enrollment
* Breast feeding
* Any current uncontrolled bacterial, fungal or viral infection

Donor:

* Pregnant, negative test must be confirmed by serum or urine pregnancy test within 14 days prior to enrollment if female
* If female, breast feeding

Max Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing grade 3-4 GVHD and/or transplant related mortality (TRM). | Within 100 days post-transplant infusion
  Safety will be measured by monitoring for the incidence of grade 3-4 GVHD as well as any transplant related mortality experience. Feasibility monitoring will include 1) failure to receive protocol directed DLI among the evaluable participants; and 2) the number of days from transplant infusion to DLI infusion among evaluable participants.

SECONDARY OUTCOMES:
Number of participants experiencing safety issues or feasibility concerns related to blinatumomab administration. | Within 180 days post-transplant infusion
  Safety and feasibility will be measured by monitoring for any early discontinuation of blinatumomab.
Describing pharmacokinetics of rabbit ATG in participants. | Within 14 days post-transplant infusion
  Measuring concentration of rabbit ATG levels in participants at the specified time points within the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Triplett, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols